CLINICAL TRIAL: NCT07208422
Title: Study Protocol for a Pilot Randomized Controlled Trial of Task-Specific Self-Rehabilitation Training (TASSRET) for Improving Functional Mobility in Community-Dwelling Stroke Survivors in a Low-Resource Setting
Brief Title: Task-Specific Self-Rehabilitation Training (TASSRET) Trial
Acronym: TASSRET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Assembly Clinic (Other)
Collaborators: Bayero University Kano, Nigeria (Other)
Responsible Party: Principal Investigator, Rabiu Ibrahim, Director of Physiotherapy, National Assembly Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: TASSRETTrial; NHREC/BUK-HREC/06/12/119/5 (Other: Bayero University Kano Health Research Ethics Committee)
Record Dates: First submitted 2025-09-27; First posted 2025-10-06 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Stroke; Stroke Hemorrhagic; Stroke Ischemic; Hemiparesis After Stroke
Keywords: Stroke rehabilitation; Task-specific Training; LMICs; Self-administered intervention; Functional ability
MeSH Terms: conditions — Stroke; Hemorrhagic Stroke; Ischemic Stroke

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Stattitician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TASSRET-video (Experimental): Participants in this group will use the TASSRET-video, which will be transferred to their phones via Xender (a file-sharing app). The application is user-friendly and features video clips of individuals demonstrating task training, accompanied by verbal explanations in Hausa. Upon opening the app, participants first view an introductory video on how to use the application. They can then navigate through three main sections: training for upper extremity function, training for lower extremity and balance function, and training for trunk strength. Each section starts with an instructional video.
  Participants will be required to select training sessions based on their rehabilitation needs, follow the videos, and perform the tasks, starting with ten repetitions or more (depending on comfort) per session. The number of repetitions is to be increased by at least 50% weekly, not exceeding a maximum of 300 repetitions per session. The training will be performed twice daily, three times per wee
  Interventions: Behavioral: Video-based Task-specific Training
- TASSRET-manual (Active Comparator): 2. TASSRET-manual: Participants in this group will be given the TASSRET-manual, which contains the same task training as the video version. The manual covers pictures of individuals demonstrating the tasks with a corresponding text description in the Hausa language. Participants will be instructed to follow the images and text descriptions to perform the tasks, mirroring the training process in the video group. The frequency, number of repetitions, and duration of the intervention are the same as in the TASSRET-video group.
  Interventions: Behavioral: Manual-based Task-specific Training

INTERVENTIONS:
Behavioral: Video-based Task-specific Training — Video-based self-administered TST
  Other Names: Video-based TST
  Arms: TASSRET-video
Behavioral: Manual-based Task-specific Training — Manual-based self-administered TST
  Other Names: Manual-based TST
  Arms: TASSRET-manual

SUMMARY:
The goal of this pilot RCT is to evaluate the effectiveness of a Task-specific Self-rehabilitation Training (TASSRET) program and compare the effect of the two formats of the TASSRET (video vs manual) on functional ability (upper extremity fine and gross motor skills, upper extremity manual dexterity and speed, voluntary movement and basic mobility, gait velocity, balance) and health-related quality of life among Hausa-native stroke survivors.

The main questions it aims to answer are:

1. What is the immediate effect and durability of TASSRET on functional ability (upper extremity fine and gross motor skills, upper extremity manual dexterity and speed, voluntary movement and basic mobility, gait velocity, balance) and health-related quality of life among the Hausa-native stroke survivors?
2. Which of the self-rehabilitation formats (TASSRET-manual or TASSRET-video) is more effective (immediate and durable) at improving functional ability (upper extremity fine and gross motor skills, upper extremity manual dexterity and speed, voluntary movement and basic mobility, gait velocity, balance) and health-related quality of life among the Hausa-native stroke survivors?

DETAILED DESCRIPTION:
Stroke is a major cause of acquired adult neurological disability worldwide, with its incidence showing a concerning upward trend in low- and middle-income countries (LMICs) over the past decade. This rise in stroke cases implies a growing burden of post-stroke disability, where functional limitations affect many survivors long-term. Approximately one-third of first-time stroke survivors may experience physical disabilities lasting five years or more, adversely impacting their community integration and quality of life. In community settings, particularly in LMICs, access to therapy and rehabilitation services is severely limited compared to hospital environments.

A recent systematic review highlighted the scarcity of high-quality, evidence-based research on rehabilitation strategies to improve functional mobility after stroke in LMICs, especially interventions that can be self-administered. Much of the existing evidence for home-based, self-administered post-stroke rehabilitation, including that based on best-practice guidelines, comes from studies in high-income countries (HICs). These models are often unsuitable for LMICs due to feasibility and affordability issues.

Another systematic review of 62 studies demonstrated that exercise-based and brain training interventions can enhance functional outcomes in LMICs post-stroke. Although techniques promoting neuroplasticity exist, task-specific training (TST) shows promise for improving outcomes in these settings. However, research on TST protocols in LMICs is limited by small sample sizes, lack of self-administration features, inadequate descriptions of exercise parameters like type, intensity, and frequency, and a focus on non-community-based settings.

To address these gaps, two formats of a task-specific self-rehabilitation training program (TASSRET-video and TASSRET-manual) were developed for use in developing countries. This protocol outlines a pilot randomized controlled trial (RCT) to investigate their effectiveness in enhancing functional mobility among community-dwelling stroke survivors.

Ethical approval was obtained from the Bayero University Kano Health Research Ethics Committee (NHREC/BUK-HREC/06/12/119/5). Permissions will be sought from community leaders, and recruitment will occur through health centers. Written consent will be obtained from all eligible participants before enrollment, in line with ethical standards.

The study employs a two-arm, outcome assessor-blinded RCT design. Participants will be randomly assigned to either the TASSRET-video or TASSRET-manual group following consent and baseline assessment. This design is chosen for its rigor in hypothesis testing and as the gold standard for evaluating intervention effectiveness.

The target population consists of Hausa-native adult stroke survivors residing in the rural communities of Kura, Karfi, and Dan Hassan in Kano State, Nigeria.

50 participants (25 per group) will be involved in this study. This was determined using G*Power software version 3.1.9.7.

Recruitment will involve community leaders identifying and introducing potential participants. Two experienced research assistants will assist in this process, collecting phone contacts and approaching individuals. Consecutive sampling will be used, enrolling eligible participants until the sample size is reached.

Following baseline data collection, participants will be randomized using block randomization. An independent statistician will generate the sequence via a computer program, excluding involvement in recruitment, treatment, or assessment. Allocation will be concealed in sequentially numbered, sealed, opaque envelopes, revealed only at assignment. Outcome assessors and data entry personnel will remain blinded to group allocation, and participants will be instructed not to disclose their group.

The interventions consist of two groups. In the TASSRET-video group, participants will receive the program via video clips transferred to their Android phones using a file-sharing application. The app includes an introductory video on usage, followed by sections on upper extremity function, lower extremity and balance function, and trunk strength. Each section begins with instructions, and participants select sessions based on needs, performing tasks while following video demonstrations with Hausa verbal explanations. They start with at least 10 repetitions per task, increasing by 50% weekly up to 300 maximum, conducted twice daily, three times per week for six weeks, preceded by warm-up exercises shown in the video.

The TASSRET-manual group will receive a printed manual with the same tasks, featuring pictures of demonstrations and Hausa text descriptions. Participants follow these to perform exercises, matching the video group's frequency, repetitions, and duration. Both groups are encouraged to involve family caregivers for assistance.

Outcomes include various measures assessed at baseline, six weeks post-intervention, and three-month follow-up. These encompass upper and lower extremity function via the Stroke Rehabilitation Assessment of Movement (STREAM), fine motor skills with the Action Research Arm Test (ARAT) and Box and Block Test (BBT), arm and hand activity using the Chedoke Arm and Hand Activity Inventory, gait with the 10-Meter Walk Test (10MWT) and 6-Minute Walk Test (6MWT), dynamic balance through the Mini-Balance Evaluation System Test (Mini-BEST), spasticity with the Modified Ashworth Scale, muscle strength using the Medical Research Council scale, quality of life via the Stroke Impact Scale (SIS), and adverse events reported by participants.

Three trained research assistants will handle assessments, each focusing on specific outcomes: one for motor skills, mobility, and adverse effects; another for dexterity, spasticity, and strength; the third for balance and gait. They will also assist in scoring the SIS for illiterate participants. Adverse events, such as discomfort or incidents, will be documented during and after intervention.

Data collection occurs at baseline (including socio-demographics and clinical info), six weeks, and three months. Each participant's data will be stored in a folder, recorded in a booklet, and entered into password-protected Microsoft Excel 2016. Hard copies will be secured. Deviations or discontinuities will be documented with reasons.

Baseline comparisons will use Mann-Whitney U or Chi-square tests of difference. Intention-to-treat with last observation carried forward will handle missing data. Repeated-measures MANOVA will examine within-subject effects, time effects, and time-by-group interactions. Univariate tests and Bonferroni-adjusted pairwise comparisons will evaluate immediate and sustained effects, with significance at p ≤ 0.05.

This pilot RCT fills a key gap in stroke rehabilitation by assessing the feasibility and initial effectiveness of self-administered TASSRET formats for community-dwelling survivors in low-resource areas. Strengths include the randomized, blinded design, validated measures, and cultural-linguistic adaptation for Hausa speakers. Comparing video and manual formats will reveal optimal delivery methods for LMICs with limited physiotherapy access.

Findings will support a larger RCT to verify TASSRET's effectiveness. The tailored approach could model scalable, affordable rehabilitation for other LMICs, improving mobility and quality of life in underserved populations.

ELIGIBILITY:
Inclusion Criteria:

* Are aged 18 years or older
* Diagnosed with a first-ever episode of ischemic or haemorrhagic stroke (including intracerebral haemorrhage and subarachnoid haemorrhage)
* Speaks and understands the Hausa language
* Living within the community and having no access to physiotherapy care
* Having access to an Android phone
* More than 10-degree extension of the index finger and abduction of the thumb
* Cognitive ability to follow commands, as indicated by a score of 0 to 1 on the Commands item of the National Institutes of Health Stroke Scale or a Mini-Mental State Examination score of ≥24
* Ability to stand and take a step (with or without support).

Exclusion Criteria:

* Had cerebrovascular events due to malignancy or head trauma
* Had been diagnosed with other neurological disorders
* Were not permanent residents of the selected communities
* Were currently receiving any form of physical rehabilitation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-06-07 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Action Research Arm Test (ARAT) | Baseline, six weeks post-intervention and three-month follow-up.
  This is a measure of upper extremity fine and gross motor skills. The scale ranges from 0 to 57, with higher scores indicating better upper extremity fine and gross motor skills.
Stroke Rehabilitation Assessment of Movement (STREAM) | Baseline, six weeks post-intervention and three-month follow-up.
  A measure of voluntary movement and basic mobility. The scale ranges from o to 100, with higher scores indicating better voluntary movement and basic mobility.
Box and Block Test (BBT) | Baseline, six weeks post-intervention and three-month follow-up.
  This measure manual dexterity and speed. The assessment is based on the number of blocks transferred from one compartment to the other within one minute. Higher scores indicate better manual dexterity and speed.
Ten-Meter Walk Test (10MWT) | Baseline, six weeks post-intervention and three-month follow-up.
  A measure of gait velocity. This is the time taken to walk a distance of ten meters, it is reported in meter per second. Lower scores indicate better gait velocity.
Mini-Balance Evaluation System Test (Mini-BEST) | Baseline, six weeks post-intervention and three-month follow-up.
  This is a measure of dynamic balance. The scores range from 0 to 28, with higher scores indicating better dynamic balance.
Stroke Impact Scale (SIS) | Baseline, six weeks post-intervention and three-month follow-up.
  A self-reported measure of health-related quality of life. The scores range from 0 to 100, with higher scores indicating better perceived health-related quality of life.

SECONDARY OUTCOMES:
Modified Ashworth scale (MAS) | Baseline, six weeks post-intervention and three-month follow-up.
  A measure of spasticity. The scores range from 0 to 4, with lower scores indicating better outcome of spasticity.
Manual Muscle Testing (MMT) | Baseline, six weeks post-intervention and three-month follow-up.
  A measure of gross muscle strength. The scores range from 0 to 5, with higher scores indicating better muscle strength.

OTHER OUTCOMES:
Adverse event | Six weeks post-intervention and three-month follow-up.
  Presence and type of adverse event.

CONTACTS AND LOCATIONS:
Overall Officials: Rabiu Ibrahim, MSc, Principal Investigator — National Assembly Clinic; Isa U Lawal, PhD, Study Chair — Bayero University Kano, Nigeria
Locations (1):
- Kura, Karfi and Dan-Hassan communities, Kano, Nigeria

IPD SHARING:
Plan to Share IPD: Yes
The results of the study will be published and be presented in scientific conferences
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: At the end of the study (sometimes in November 2025)
Access Criteria: The Raw data (anonymized) can be accessed from the principal investigator on request.

REFERENCES:
- [Background] Ibrahim R, Joseph C, Stewart A, Lawal IU. Self-rehabilitation strategy for rural community-dwelling stroke survivors in a lower-middle income country: a modified Delphi study. PLoS One. 2025 Feb 25;20(2):e0303658. doi: 10.1371/journal.pone.0303658. eCollection 2025. PMID 39999052
- See also: The article reported the development of the Task-specific Self-rehabilitation intervention (TASSRET). This protocol described how the effectiveness of two formats of this intervention will be evaluated via pilot RCT — https://doi.org/10.1371/journal.pone.0303658